CLINICAL TRIAL: NCT03784183
Title: A Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy of a Non-Pharmacological Intervention of Cognitive Stimulation in Subjects With Alzheimer's Disease and Mild Cognitive Impairment: The Brain Stimulation Project.
Brief Title: Neuropsychological and Neurophysiological Effects of Cognitive Stimulation in Patients With Alzheimer's Disease and Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Carlo de Lena, Department of Human Neuroscience, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSP-2018
Record Dates: First submitted 2018-11-26; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Mild Cognitive Stimulation; Non Pharmacological Intervention; Cognitive Stimulation; Transcranial Magnetic Stimulation; Blink Reflex; Neuropsychological Evaluation; Randomized Controlled Trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A Randomized, Single-Blind, Placebo-Controlled, Parallel-Group
Who Masked: Outcomes Assessor
Masking Description: Single Blind: Neuropsychologists and Neurophysiologists are prevented from having knowledge of the intervention assigned to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- moderate AD-experimental (Experimental): Experimental Intervention: The CS shall be carried out in groups (5-7 participants), twice a week. Each session lasts 90 minutes. CS sessions begin with a training for temporal and spatial orientation in which participants are asked to recognize and recall the date and the place with the help of some environmental aids (calendars, clocks, pictures and maps). Then the participants complete an array of cognitive tasks for memory, attention, language, visuo-spatial functions and executive functions. These tasks range from individual paper-and-pencil exercises to verbal-learning exercises that have to be solved by the group.
  Interventions: Other: Cognitive Stimulation (CS)
- mild AD-experimental (Experimental): Experimental Intervention: the same of the "moderate AD-experimental" arm
  Interventions: Other: Cognitive Stimulation (CS)
- MCI-experimental (Experimental): Experimental Intervention: the same of the "moderate AD-experimental" arm
  Interventions: Other: Cognitive Stimulation (CS)
- moderate AD-placebo (No Intervention)
- mild AD-placebo (No Intervention)
- MCI-placebo (No Intervention)

INTERVENTIONS:
Other: Cognitive Stimulation (CS) — CS consists of a wide range of structured activities aimed at the general improvement of social functioning and the maintenance of different cognitive functions. It is a non-specific in-group approach that places particular emphasis on social interactions.
  Arms: MCI-experimental; mild AD-experimental; moderate AD-experimental

SUMMARY:
The present study aims to evaluate the effect of cognitive stimulation (CS) in participants with a diagnosis of moderate and mild Alzheimer's disease (AD) and mild cognitive impairment (MCI) compared to control subjects not receiving any non-pharmacological interventions. Treated participants will receive a structured CS consisting of a wide range of activities aimed at the general improvement of social functioning and the maintenance of cognitive functions. The study consists of a 24-week treatment phase and a follow-up period of 24 weeks. During the treatment period, patients will receive two CS sessions a week. At baseline, all the participants undergo an extensive neuropsychological evaluation and a neurophysiological assessment aimed at studying the frequency of spontaneous blinking (blink rate) and cortical excitability and synaptic plasticity by means of the transcranial magnetic stimulation (TMS). Neuropsychological and neurophysiological evaluations will be repeated at the end of the treatment (week 24) and at the end of the follow-up period (week 48) in order to evaluate short- and long-term effects of CS. The hypothesis of this research is that CS may improve cognition and the neurophysiological parameters studied in treated participants compared to those untreated.

ELIGIBILITY:
Inclusion Criteria:

1. moderate AD participants

   * Clinical diagnosis of probable AD (National Institute on Aging and Alzheimer's Association criteria)
   * 1 < Clinical Dementia Rating Scale < 3
   * 13 ≤ Mini-Mental State Examination < 20/30
   * Modified Hachinski Ischaemic Scale (MHIS) ≤ 4
   * Geriatric Depression Scale (GDS) ≤ 6
2. mild AD participants

   * Clinical diagnosis of probable AD (National Institute on Aging and Alzheimer's Association criteria)
   * Clinical Dementia Rating Scale = 1 (memory box score ≥ 0.5)
   * 20 > Mini-Mental State Examination < 27/30
   * Modified Hachinski Ischaemic Scale (MHIS) ≤ 4
   * Geriatric Depression Scale (GDS) ≤ 6
3. MCI participants

   * Clinical diagnosis of probable AD (National Institute on Aging and Alzheimer's Association criteria)
   * Clinical Dementia Rating Scale < 1 (memory box score ≥ 0.5)
   * Mini-Mental State Examination ≥ 24/30
   * Modified Hachinski Ischaemic Scale (MHIS) ≤ 4
   * Geriatric Depression Scale (GDS) ≤ 6

Exclusion Criteria for all the participants (moderate AD, mild AD and MCI):

* Any medical or neurological condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause of the subject's cognitive impairment.
* Clinically significant psychiatric illness (e.g., uncontrolled major depression, bipolar affective disorder) within 6 months prior to the enrolment.
* Any medications that, in the opinion of the Investigator, may contribute to cognitive impairment or impair the subject's ability to perform cognitive testing or complete study procedures.
* Contraindications to Transcranial Magnetic Stimulation (history of epilepsy or seizures/presence of pacemaker).
* Subject currently living in an organized care facility with extensive intervention and/or support of daily living activities.
* Inability to comply with study requirements and commitments
* Has not one informant/care partner who, in the Investigator's opinion, has frequent and sufficient contact with the subject as to be able to provide accurate information about the subject's cognitive and functional abilities.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in global cognition as assessed by Mini Mental State Examination | 24 and 48 weeks
  Change from baseline in Mini Mental State Examination score at Week 24 and 48. This scale investigates global cognition. Scale range: 0-30. Normal values >24. Higher values represent a better outcome.
Change in dementia severity as assessed by Clinical Dementia Rating Scale | 24 and 48 weeks
  Change from baseline in Clinical Dementia Rating Scale score at Week 24 and 48. This scale investigates global cognition and dementia severity. Scale range: 0-5. Normal values = 0. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Change in frontal functions as assessed by Frontal Assessment Battery | 24 and 48 weeks
  Change from baseline in Frontal Assessment Battery scores at Week 24 and 48. This scale investigates the executive functions. Scale range: 0-30. Normal values ≥ 13.5. Higher values represent a better outcome.
Change in verbal memory as assessed by Rey Auditory Verbal Learning Test | 24 and 48 weeks
  Change from baseline in Rey Auditory Verbal Learning Test scores at Week 24 and 48. This test investigates verbal learning and memory. Immediate recall scale range: 0-75. Normal values >28.52. Delayed recall scale range: 0-15. Normal values >4.68. Higher values represent a better outcome.
Change in attention as assessed by Visual Search Test | 24 and 48 weeks
  Change from baseline in Visual Search test score at Week 24 and 48. This test investigates selective attention. Scale range: 0-60. Normal values >30. Higher values represent a better outcome.
Change in visuospatial functions as assessed by Clock Drawing Test | 24 and 48 weeks
  Change from baseline in Clock Drawing Test score at Week 24 and 48. This test investigates visuospatial abilities and executive functioning. Scale range: 0-61. Normal values >42.17. Higher values represent a better outcome.
Change in naming as assessed by Boston Naming Test | 24 and 48 weeks
  Change from baseline in Boston Naming test score at Week 24 and 48. This test measure object naming from line drawings. Scale range: 0-60. Normal values >24. Higher values represent a better outcome.
Change in synaptic plasticity as assessed by Paired Associative Stimulation | 24 and 48 weeks
  Change from baseline in Paired Associative Stimulation at Week 24 and 48. Paired associative stimulation is a paradigm combining peripheral nerve stimulation and transcranial magnetic stimulation over the contralateral primary motor cortex. In healthy humans, Paired Associative Stimulation after-effects last about 30-60 minutes. The extent of facilitatory-Paired Associative Stimulation-induced effects on MEP amplitude ranges from 120% to 160%, while inhibitory-Paired Associative Stimulation may induce a reduction of muscle-evoked potential amplitude that ranges from 60% to 90%.
Change in blinking as assessed by Blink Rate Evaluation | 24 and 48 weeks
  Change from baseline in the blink rate at Week 24 and 48. Spontaneous blinking was measured by the Blink Rate and was expressed as number of blinks per minute. Normal values: mean Blink Reflex value at rest is 17 blinks/minute; during conversation is 26 blinks/minute; during reading is 4.5 blinks/minute. Cut offs: not applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Neuroscience, Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided